CLINICAL TRIAL: NCT03339206
Title: Enhancing Source Credibility in Tobacco Regulatory Communications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Goldstein, MD, MPH, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-0610; P50CA180907 (NIH)
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Cigarette Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking | interventions — United States Food and Drug Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Constituent message with FDA and quitline (Experimental): Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm will also include an FDA logo, and information about the benefits of quitting smoking and the quitline. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Interventions: Behavioral: Constituent message with FDA and quitline
- Constituent message without FDA and quitline (Experimental): Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm is identical to the arm above, except that it does not include FDA source or quit information. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Interventions: Behavioral: Constituent message without FDA and quitline
- Littering message (Control) (Other): Messages about littering cigarettes will include text designed to discourage people from littering their cigarette butts, and an image related to the message. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Interventions: Behavioral: Littering message (Control)

INTERVENTIONS:
Behavioral: Constituent message with FDA and quitline — Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm will also include an FDA logo, and information about the benefits of quitting smoking and the quitline. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Arms: Constituent message with FDA and quitline
Behavioral: Constituent message without FDA and quitline — Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm is identical to the arm above, except that it does not include FDA source or quit information. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Arms: Constituent message without FDA and quitline
Behavioral: Littering message (Control) — Messages about littering cigarettes will include text designed to discourage people from littering their cigarette butts, and an image related to the message. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators used text developed by investigators associated with our Center for Regulatory Research on Tobacco Communication. Design of these messages was developed by our team.
  Arms: Littering message (Control)

SUMMARY:
This study will assess the impact of cigarette constituent messages with and without FDA source and quit information in a randomized controlled trial. The investigators hypothesize that cigarette constituent messages will increase intention to quit compared to messages about littering cigarettes (the control). The investigators also hypothesize that constituent messages that include FDA source and quit information will increase intention to quit compared to messages without that information.

DETAILED DESCRIPTION:
The Family Smoking Prevention and Tobacco Control Act delegates the U.S. Food and Drug Administration (FDA) to communicate the risks of smoking to the public, among other tobacco regulatory responsibilities. Little research exists about how FDA, as a regulatory agency, should develop and deliver these messages, and whether they should include their source information on the ads. This study will assess the impact of cigarette constituent messages with and without FDA source and quit information in a randomized controlled trial.

Recruitment: People interested in participating will complete an online screener. Study staff will invite people eligible based on the screener to enroll in the study.

Informed Consent: The consent form will be shared with people who are eligible based on the screener in the invitation email. At the beginning of the baseline survey, participants will again review the consent form and will be asked to provide consent in order to enroll in the study.

Randomization: At the end of the baseline survey, survey software will randomly assign participants to one of the three study arms. Participants will have an equal chance of being randomized to each study arm.

Assessment: Participants will complete 18 computer based surveys during the study. The first baseline survey will take around 20 minutes to complete on day 0. Participants will then receive a survey each morning for days 1-15 that will include behavior measures as well as their assigned study intervention. These surveys will take approximately 5 minutes to complete. Participants will then complete a 20-minute survey on day 16, and day 32.

Detailed description of the intervention: Participants will receive an email with a link to a survey each morning for 15 days. During that survey they will be shown one message from their condition. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order. Study investigators designed the messages.

ELIGIBILITY:
Inclusion Criteria:

* Have smoked at least 100 cigarettes in his or her lifetime
* Currently smoke cigarettes every day or some days
* Work or home access to the internet
* Email account that is regularly used
* Lives in the US
* Comfortable taking a survey in English
* Able to complete a survey on a computer
* Able to complete surveys delivered via email
* Able to complete 3, 20 minute surveys during the study
* Able to complete surveys in the morning for 15 days

Exclusion Criteria:

* Currently using pharmacotherapy, a quitline, or a quit smoking program or support group for smoking cessation
* Participated in a research study about smoking cigarettes or using other tobacco products in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 845 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Goldstein AO, Jarman KL, Kowitt SD, Queen TL, Kim KS, Shook-Sa BE, Sheeran P, Noar SM, Ranney LM. Effect of Cigarette Constituent Messages With Engagement Text on Intention to Quit Smoking Among Adults Who Smoke Cigarettes: A Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210045. doi: 10.1001/jamanetworkopen.2021.0045. PMID 33625509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and screened for study eligiblity online between June 2017 and April 2018, and invited to enroll after the study started and they were determined to be eligible.
Pre-assignment Details: 845 participants consented to participate in the study, of those 41 did not complete the baseline questionnaire and were not randomized. Of the 804 originally reported 12 were ineligible since they were not current smokers, 1 person withdrew, and 2 were duplicates. Our final analytic sample is 789.
Groups:
- Constituent Message With FDA and Quitline: Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm will also include an FDA logo, and information about the benefits of quitting smoking and the quitline. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order.
  Constituent message with FDA and quitline: Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm will also include an FDA logo, and information about the benefits of quitting smoking and the quitline. Each condition has 5 messages that will be r
- Constituent Message Without FDA and Quitline: Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm is identical to the arm above, except that it does not include FDA source or quit information. Each condition has 5 messages that will be repeated 3 times in a counterbalanced order.
  Constituent message without FDA and quitline: Messages about the chemical constituents of cigarette smoke will include text about chemicals in cigarette smoke and health effects of the chemicals, and an image of a person related to the health effect. This arm is identical to the arm above, except that it does not include FDA source or quit information. Each condition has 5 messages that will be repeated 3 times
Period: Overall Study
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Started | 262 | 263 | 264
Completed | 262 | 263 | 264
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control) | Total
Number analyzed (Participants) | 262 | 263 | 264 | 789
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants who responded to the measure at the time point of interest
  years
    number analyzed (Participants) | 261 | 262 | 264 | 787
    (all) | 43.95 (12.88) | 42.83 (12.71) | 43.33 (13.08) | 43.37 (12.88)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 99 | 96 | 106 | 301
  Female | 161 | 166 | 156 | 483
  Gender non-conforming | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 27 | 23 | 72
  Not Hispanic or Latino | 240 | 236 | 241 | 717
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 192 | 181 | 205 | 578
  Black or African American | 52 | 63 | 49 | 164
  Other Race | 18 | 19 | 10 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 262 | 263 | 264 | 789

OUTCOME MEASURES:

1. Primary Outcome: Quit Intentions
Description: Average quit intention score measured at 16 days by survey. Quit intention measured with 3 questions, the final quit intention score is a mean of the response to the 3 questions, on a scale of 1 to 4, where 1 indicates low intention to quit, and 4 indicates a high intention to quit.
Time Frame: day 16
Population: Participants who responded to the measure at the time point of interest, post 1 (day 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 232 | 228
score on a scale | 2.73 (0.95) | 2.67 (0.94) | 2.58 (1.00)

2. Secondary Outcome: Number of Cigarettes Smoked Each Day
Description: Measured daily by survey
Time Frame: days 1-15
Population: Overall number of participants analyzed is the number of participants in each condition that responded to the outcome measure for at least one time point. Participants who responded to the measure at the time point of interest are included in the row for that time point, but participants that did not are excluded for that day.
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked each day
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 234 | 237
Number of cigarettes smoked each day
  Day 1: number analyzed (Participants) | 173 | 174 | 176
  Day 1 | 15.06 (9.16) | 14.16 (9.78) | 15.77 (10.14)
  Day 2: number analyzed (Participants) | 189 | 185 | 188
  Day 2 | 15.79 (10.39) | 14.67 (11.34) | 15.94 (9.82)
  Day 3: number analyzed (Participants) | 190 | 190 | 187
  Day 3 | 15.41 (10.61) | 13.59 (9.05) | 14.27 (8.58)
  Day 4: number analyzed (Participants) | 186 | 181 | 192
  Day 4 | 15.00 (10.24) | 13.85 (9.69) | 14.59 (8.69)
  Day 5: number analyzed (Participants) | 187 | 199 | 185
  Day 5 | 14.35 (9.80) | 13.52 (8.44) | 14.56 (9.67)
  Day 6: number analyzed (Participants) | 178 | 188 | 183
  Day 6 | 14.15 (10.42) | 13.64 (10.41) | 13.60 (9.56)
  Day 7: number analyzed (Participants) | 178 | 181 | 165
  Day 7 | 13.91 (10.17) | 13.13 (10.08) | 13.64 (8.99)
  Day 8: number analyzed (Participants) | 185 | 196 | 183
  Day 8 | 13.98 (9.93) | 13.14 (10.15) | 13.37 (9.00)
  Day 9: number analyzed (Participants) | 186 | 193 | 182
  Day 9 | 14.40 (10.97) | 12.94 (9.47) | 13.74 (9.93)
  Day 10: number analyzed (Participants) | 184 | 187 | 173
  Day 10 | 14.15 (10.66) | 12.29 (9.68) | 13.51 (8.75)
  Day 11: number analyzed (Participants) | 187 | 195 | 189
  Day 11 | 14.24 (10.24) | 12.84 (9.46) | 13.40 (9.16)
  Day 12: number analyzed (Participants) | 199 | 198 | 189
  Day 12 | 14.09 (10.22) | 12.83 (9.56) | 13.57 (9.37)
  Day 13: number analyzed (Participants) | 198 | 199 | 201
  Day 13 | 14.23 (9.76) | 12.67 (9.80) | 13.25 (9.10)
  Day 14: number analyzed (Participants) | 187 | 192 | 184
  Day 14 | 14.53 (10.64) | 12.64 (9.37) | 13.87 (9.16)
  Day 15: number analyzed (Participants) | 200 | 197 | 185
  Day 15 | 13.75 (10.09) | 11.92 (8.69) | 13.65 (8.63)

3. Secondary Outcome: Number of Cigarettes Forgone Each Day
Description: Measured daily by survey
Time Frame: days 1-15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of cigarettes forgone each day
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 234 | 237
Number of cigarettes forgone each day
  Day 1: number analyzed (Participants) | 173 | 175 | 176
  Day 1 | 1.08 (1.87) | 0.91 (1.20) | 1.30 (2.10)
  Day 2: number analyzed (Participants) | 189 | 185 | 188
  Day 2 | 1.11 (1.53) | 1.12 (1.48) | 1.29 (1.82)
  Day 3: number analyzed (Participants) | 192 | 190 | 187
  Day 3 | 1.22 (1.70) | 1.38 (1.72) | 1.37 (2.17)
  Day 4: number analyzed (Participants) | 187 | 181 | 192
  Day 4 | 1.39 (1.97) | 1.30 (1.52) | 1.66 (3.90)
  Day 5: number analyzed (Participants) | 187 | 199 | 185
  Day 5 | 2.05 (7.57) | 1.43 (2.35) | 1.83 (7.54)
  Day 6: number analyzed (Participants) | 179 | 188 | 183
  Day 6 | 2.24 (7.72) | 1.35 (1.66) | 1.40 (2.33)
  Day 7: number analyzed (Participants) | 179 | 181 | 166
  Day 7 | 1.68 (2.34) | 1.53 (1.92) | 1.52 (2.10)
  Day 8: number analyzed (Participants) | 185 | 196 | 183
  Day 8 | 2.15 (7.61) | 1.61 (2.01) | 1.48 (2.31)
  Day 9: number analyzed (Participants) | 187 | 193 | 182
  Day 9 | 2.17 (7.53) | 1.40 (1.83) | 1.55 (2.61)
  Day 10: number analyzed (Participants) | 184 | 187 | 173
  Day 10 | 2.12 (7.67) | 1.40 (1.89) | 1.62 (2.62)
  Day 11: number analyzed (Participants) | 187 | 195 | 189
  Day 11 | 1.94 (7.57) | 1.46 (1.79) | 1.63 (2.36)
  Day 12: number analyzed (Participants) | 200 | 198 | 190
  Day 12 | 1.89 (7.30) | 1.55 (2.01) | 1.63 (2.53)
  Day 13: number analyzed (Participants) | 198 | 199 | 201
  Day 13 | 1.92 (7.36) | 1.36 (1.86) | 1.42 (2.22)
  Day 14: number analyzed (Participants) | 187 | 193 | 184
  Day 14 | 1.42 (2.07) | 1.38 (1.60) | 1.57 (2.29)
  Day 15: number analyzed (Participants) | 200 | 197 | 186
  Day 15 | 2.00 (7.31) | 1.53 (1.97) | 1.52 (2.68)

4. Secondary Outcome: Number of Cigarettes Butted Out Each Day
Description: Measured daily by survey
Time Frame: days 1-15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of cigarettes butted out per day
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 234 | 237
Number of cigarettes butted out per day
  Day 1: number analyzed (Participants) | 173 | 175 | 176
  Day 1 | 1.42 (2.28) | 1.53 (2.10) | 1.91 (3.12)
  Day 2: number analyzed (Participants) | 189 | 185 | 188
  Day 2 | 1.69 (2.78) | 1.44 (2.21) | 2.11 (3.64)
  Day 3: number analyzed (Participants) | 192 | 190 | 187
  Day 3 | 1.72 (2.60) | 1.49 (2.04) | 1.71 (2.60)
  Day 4: number analyzed (Participants) | 187 | 181 | 192
  Day 4 | 1.72 (2.59) | 1.59 (2.09) | 2.15 (4.34)
  Day 5: number analyzed (Participants) | 187 | 199 | 185
  Day 5 | 2.28 (7.66) | 1.63 (2.04) | 1.99 (3.73)
  Day 6: number analyzed (Participants) | 179 | 188 | 183
  Day 6 | 1.89 (3.19) | 1.54 (2.03) | 1.88 (3.68)
  Day 7: number analyzed (Participants) | 179 | 181 | 166
  Day 7 | 1.72 (2.88) | 1.55 (2.04) | 1.87 (3.44)
  Day 8: number analyzed (Participants) | 185 | 196 | 183
  Day 8 | 2.26 (7.71) | 1.62 (2.11) | 1.95 (3.35)
  Day 9: number analyzed (Participants) | 187 | 193 | 182
  Day 9 | 2.12 (7.65) | 1.57 (2.15) | 1.81 (3.34)
  Day 10: number analyzed (Participants) | 184 | 187 | 173
  Day 10 | 2.15 (7.75) | 1.22 (1.68) | 2.16 (3.86)
  Day 11: number analyzed (Participants) | 187 | 195 | 189
  Day 11 | 2.19 (7.69) | 1.43 (1.93) | 2.07 (3.70)
  Day 12: number analyzed (Participants) | 200 | 198 | 190
  Day 12 | 2.04 (7.46) | 1.44 (2.05) | 1.95 (3.41)
  Day 13: number analyzed (Participants) | 198 | 199 | 201
  Day 13 | 2.06 (7.52) | 1.36 (1.98) | 1.82 (3.25)
  Day 14: number analyzed (Participants) | 187 | 193 | 184
  Day 14 | 1.59 (2.26) | 1.57 (2.14) | 2.01 (3.45)
  Day 15: number analyzed (Participants) | 200 | 197 | 186
  Day 15 | 2.11 (7.45) | 1.51 (2.27) | 1.84 (3.38)

5. Secondary Outcome: Quit Attempts During the Study
Description: Measured by survey
Time Frame: days 16 and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 236 | 242 | 236
Participants
  Made Quit Attempt as of Post 1 (day 16): number analyzed (Participants) | 232 | 232 | 229
  Made Quit Attempt as of Post 1 (day 16) | 58 | 59 | 51
  Made Quit Attempt as of Post 2 (day 32): number analyzed (Participants) | 227 | 233 | 228
  Made Quit Attempt as of Post 2 (day 32) | 90 | 99 | 105

6. Secondary Outcome: Awareness of Quitline
Description: Measured by survey
Time Frame: day 16
Population: Participants who responded to the measure at the time point of interest, post 1 (day 16)
Measure: Count of Participants; unit: Participants
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 232 | 229
Participants
  Aware of Quitline | 122 | 107 | 95
  Not Aware of Quitline | 110 | 125 | 134

7. Secondary Outcome: Recall of Quitline Phone Number
Description: Measured by survey
Time Frame: day 16
Population: Participants who responded to the measure at the time point of interest, post 1 (day 16)
Measure: Count of Participants; unit: Participants
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 232 | 232 | 229
Participants
  Correctly recalled Quitline phone number | 70 | 45 | 49
  Did not correctly recall Quitline phone number | 162 | 187 | 180

8. Secondary Outcome: Use of Quitline During the Study
Description: Measured by survey
Time Frame: days 16 and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 236 | 242 | 236
Participants
  Reported calling Quitline at post 1 (day 16): number analyzed (Participants) | 232 | 232 | 228
  Reported calling Quitline at post 1 (day 16) | 9 | 7 | 8
  Reported calling Quitline at post 2 (day 32): number analyzed (Participants) | 227 | 233 | 228
  Reported calling Quitline at post 2 (day 32) | 23 | 21 | 16

9. Secondary Outcome: Intention to Use the Quitline
Description: Measured by survey. Intention to use the quitline was measured with one item on a 1 to 4 scale, where 1 indicates a low likelihood of calling the quitline, and 4 indicates a high likelihood of calling the quitline.
Time Frame: days 16 and 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 236 | 242 | 236
units on a scale
  Post 1 (day 16): number analyzed (Participants) | 232 | 232 | 227
  Post 1 (day 16) | 2.34 (1.14) | 2.25 (1.09) | 2.18 (1.10)
  Post 2 (day 32): number analyzed (Participants) | 227 | 233 | 228
  Post 2 (day 32) | 2.42 (1.14) | 2.29 (1.09) | 2.10 (1.12)

10. Secondary Outcome: Quit Intentions
Description: Average quit intention score measured at 32 days by survey. Quit intention measured with 3 questions, the final quit intention score is a mean of the response to the 3 questions, on a scale of 1 to 4, where 1 indicates low intention to quit, and 4 indicates a high intention to quit.
Time Frame: day 32
Population: Participants who responded to the measure at the time point of interest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 227 | 233 | 228
score on a scale | 2.78 (0.97) | 2.76 (0.97) | 2.73 (1.01)

11. Secondary Outcome: Self Efficacy
Description: Measured by survey. Self efficacy measured with 1 question, on a scale of 1 to 5, where 1 indicates low self efficacy to quit, and 5 indicates a high self efficacy to quit smoking cigarettes.
Time Frame: days 16 and 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 236 | 241 | 236
units on a scale
  Post 1 (Day 16): number analyzed (Participants) | 232 | 231 | 227
  Post 1 (Day 16) | 2.83 (1.13) | 2.84 (1.08) | 2.69 (1.10)
  Post 2 (Day 32): number analyzed (Participants) | 227 | 233 | 228
  Post 2 (Day 32) | 2.98 (1.23) | 2.95 (1.18) | 2.89 (1.11)

12. Secondary Outcome: Response Efficacy
Description: Measured by survey. Response efficacy measured with 1 question, on a scale of 1 to 5, where 1 indicates low response efficacy of quitting, and 5 indicates a high response efficacy of quitting smoking cigarettes.
Time Frame: days 16 and 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
Number analyzed (Participants) | 236 | 241 | 236
units on a scale
  Post 1 (day 16): number analyzed (Participants) | 232 | 231 | 227
  Post 1 (day 16) | 4.24 (0.96) | 4.26 (0.97) | 4.31 (0.96)
  Post 2 (day 32): number analyzed (Participants) | 227 | 233 | 228
  Post 2 (day 32) | 4.40 (0.90) | 4.36 (0.96) | 4.36 (0.98)

ADVERSE EVENTS:
Time Frame: Low risk study, no adverse event data collected
Description: Low risk study, no adverse event data collected
Arm/Group | Constituent Message With FDA and Quitline | Constituent Message Without FDA and Quitline | Littering Message (Control)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT03339206/Prot_SAP_ICF_000.pdf